CLINICAL TRIAL: NCT06696924
Title: Comparative Effects of Reciprocal Inhibition and Static Stretching on Serratus Anterior Muscle on Pain, Range of Motion and Functional Ability Among Female Amateur Athletes.
Brief Title: Comparitive Effects of Reciprocal Inhibtion and Static Stretching Among Female Athletes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR and AHS/24/0412
Record Dates: First submitted 2024-11-18; First posted 2024-11-20 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Sports Physical Therapy
Keywords: Reciprocal inhibition; Static stretching; Serratus Anterior
MeSH Terms: interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reciprocal inhibition (Experimental): First Subjects will start doing baseline warmup exercises which are mentioned then they will perform reciprocal inhibition of the serratus muscle in side-lying. After identifying the antagonist muscles of the serratus anterior, which are typically the rhomboids or the middle and lower trapezius. Athletes will perform a gentle contraction of the antagonist's muscles by retracting or squeezing their shoulder blades together. While the antagonist muscles are contracting, we will ask the athlete to simultaneously relax and lengthen the serratus anterior muscle. The patient can achieve this by protracting or pushing their shoulder blades forward and away from each other.
  Interventions: Other: Reciprocal inhibition
- Static Stretching (Experimental): After performing baseline warmup exercises, Athlete will perform 2 exercises Standing wall stretch and seated cross body stretch
  Interventions: Other: Static stretching

INTERVENTIONS:
Other: Reciprocal inhibition — First Subjects will start doing baseline warmup exercises which are mentioned then they will perform reciprocal inhibition of the serratus muscle in supine or side-lying. After identifying the antagonist muscles of the serratus anterior, which are typically the rhomboids or the middle and lower trapezius. Athletes will perform a gentle contraction of the antagonist's muscles by retracting or squeezing their shoulder blades together. While the antagonist muscles are contracting, we will ask the athlete to simultaneously relax and lengthen the serratus anterior muscle. The patient can achieve this by protracting or pushing their shoulder blades forward and away from each other.
  Arms: Reciprocal inhibition
Other: Static stretching — Subjects will perform 2 stretches
  1. Standing Wall Stretch: Stand facing a wall with your feet about hip-width apart. Place their palms on the wall at shoulder height, slightly wider than shoulder-width apart. will Lean their body forward, keeping their arms straight, until feel a stretch in their serratus anterior. Hold the stretch for 15 to 30 seconds, then slowly release. Instead of using a wall or object, the athlete will use their opposite hand to hold the stretched arm in position.
  2. Seated Cross-Body Stretch: Sit on the edge of a chair or bench. Cross one arm over your chest, placing your hand on the opposite shoulder. The athlete will use the other hand to gently pull the crossed arm closer to your body, feeling a stretch in the serratus anterior. Hold the stretch for 15 to 30 seconds or more, and then switch sides and repeat.
  Arms: Static Stretching

SUMMARY:
The aim of the study is to determine the Comparative effects of Reciprocal Inhibition and Static Stretching on Serratus anterior Muscle on Pain, range of Motion, and Functional ability among Female Amateur Athletes

DETAILED DESCRIPTION:
There is an absence of extensive studies comparing the effects of reciprocal inhibition and static stretching specifically on the serratus anterior muscle among female amateur athletes. While some research exists on the general effects of these techniques, there is a gap in gender-specific studies and their application to amateur athletes. By conducting more detailed research in this area, we can better understand how these affect athletes, their pain levels, range of motion, and overall functional ability. This would provide valuable insights for designing warm-up routines and optimizing performance for female amateur athletes.

ELIGIBILITY:
Inclusion Criteria:

* Females
* Ages between 17-30 years
* Amateur athletes ( badminton, weight lifting, Volleyball, tennis)
* Pain in the upper limb ( Moderate pain 5-6 level on NPRS scale)
* To check Serratus anterior ( females with strength test positive and shakiness weakness on pressing or overhead activities )
* Overhead range of motion of the shoulder ( those with less than 180 degrees)

Exclusion Criteria:

* Fractures
* Musculoskeletal problems ( radiculopathy, myelopathy, inflammatory arthritis)
* International athletes
* Recent surgery thoracic spine

Ages: 17 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 56 (Actual)
Dates: Start 2024-05-24 (Actual); Primary Completion 2025-02-15 (Estimated); Study Completion 2025-02-20 (Estimated)

PRIMARY OUTCOMES:
Pain scale | 6 weeks
  For measuring pain, the Numeric Pain Rating Scale (NPRS) will be used. The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable"). This will be asked prior to exercise and after 6 weeks .
Range of motion | 6 weeks
  It will be assessed using a goniometer for the shoulder before starting the exercises and after 6 weeks.
Upper Extremity Functional Scale | 6 weeks
  It is a questionnaire related to daily activities which are asked by athletes who have upper extremity issues to check in which activity they are facing issues.

CONTACTS AND LOCATIONS:
Overall Officials: Areeza hamid, DPT, Principal Investigator — Riphah International University
Locations (1):
- Pakistan Sports Board, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barcia AM, Makovicka JL; MRAB Study Group; Spenciner DB, Chamberlain AM, Jacofsky MC, Gabriel SM, Moroder P, von Rechenberg B, Sengun MZ, Tokish JM. Scapular motion in the presence of rotator cuff tears: a systematic review. J Shoulder Elbow Surg. 2021 Jul;30(7):1679-1692. doi: 10.1016/j.jse.2020.12.012. Epub 2021 Feb 2. PMID 33540119
- [Background] Arntz F, Markov A, Behm DG, Behrens M, Negra Y, Nakamura M, Moran J, Chaabene H. Chronic Effects of Static Stretching Exercises on Muscle Strength and Power in Healthy Individuals Across the Lifespan: A Systematic Review with Multi-level Meta-analysis. Sports Med. 2023 Mar;53(3):723-745. doi: 10.1007/s40279-022-01806-9. Epub 2023 Jan 31. PMID 36719536
- [Background] Xu X, Lin JH, McGorry RW. A regression-based 3-D shoulder rhythm. J Biomech. 2014 Mar 21;47(5):1206-10. doi: 10.1016/j.jbiomech.2014.01.043. Epub 2014 Jan 30. PMID 24534377
- [Background] Wagner ER, Hussain ZB, Karzon AL, Warner JJP, Elhassan BT, Sanchez-Sotelo J. The Scapula: The Greater Masquerader of Shoulder Pathologies. Instr Course Lect. 2024;73:587-607. PMID 38090927
- [Background] Gillani SN, Ain Q-, Rehman SU, Masood T. Effects of eccentric muscle energy technique versus static stretching exercises in the management of cervical dysfunction in upper cross syndrome: a randomized control trial. J Pak Med Assoc. 2020 Mar;70(3):394-398. doi: 10.5455/JPMA.300417. PMID 32207413
- [Background] Osama M, Shakil Ur Rehman S. Effects of static stretching as compared to autogenic inhibition and reciprocal inhibition muscle energy techniques in the management of mechanical neck pain: a randomized controlled trial. J Pak Med Assoc. 2020 May;70(5):786-790. doi: 10.5455/JPMA.9596. PMID 32400728
- [Background] Jawade S, Chitale N Jr, Phansopkar P. The Effect of Reciprocal Inhibition Techniques on Pain, Range of Motion, and Functional Activities in Patients With Upper Trapezitis. Cureus. 2023 Feb 1;15(2):e34487. doi: 10.7759/cureus.34487. eCollection 2023 Feb. PMID 36874329
- [Background] Joshi R, Poojary N. The Effect of Muscle Energy Technique and Posture Correction Exercises on Pain and Function in Patients with Non-specific Chronic Neck Pain Having Forward Head Posture-a Randomized Controlled Trail. Int J Ther Massage Bodywork. 2022 Jun 1;15(2):14-21. doi: 10.3822/ijtmb.v15i2.673. eCollection 2022 Jun. PMID 35686175
- [Background] Hsu FY, Tsai KL, Lee CL, Chang WD, Chang NJ. Effects of Dynamic Stretching Combined With Static Stretching, Foam Rolling, or Vibration Rolling as a Warm-Up Exercise on Athletic Performance in Elite Table Tennis Players. J Sport Rehabil. 2020 Apr 28;30(2):198-205. doi: 10.1123/jsr.2019-0442. PMID 32350145
- [Background] Zeleznik P, Jelen A, Kalc K, Behm DG, Kozinc Z. Acute effects of static and proprioceptive neuromuscular facilitation stretching on hamstrings muscle stiffness and range of motion: a randomized cross-over study. Eur J Appl Physiol. 2024 Mar;124(3):1005-1014. doi: 10.1007/s00421-023-05325-x. Epub 2023 Oct 6. PMID 37803178